CLINICAL TRIAL: NCT01068093
Title: Assessment of the Effects of Ezetimibe on Coronary Plaque Volume in Patients With Acute Coronary Syndrome
Brief Title: The Effects of Ezetimibe on Coronary Plaque Volume in Patients With Acute Coronary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yokohama City University Medical Center (Other)
Responsible Party: Kiyoshi Hibi, Yokohama City University Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-ACS-E
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ezetimibe — 10mg daily

SUMMARY:
The purpose of this study is to assess the effects of Ezetimibe on coronary plaque volume in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
Previous studies reported that administration of statins in patients with coronary artery disease resulted in significant reduction of low-density lipoprotein cholesterol(LDL-C) and regression of coronary plaque volume, and a decrease in the level of LDL-C through statin treatment positively correlates with a reduction in the volume of plaques. Administration of Ezetimibe in addition to statin has been shown to be more effective at reducing LDL-C levels compared with statin monotherapy. However, the effects of Ezetimib on coronary plaque volume remain unclear. In this study, the investigators assess the effect of Ezetimibe on coronary plaque volume and tissue composition in patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed as acute coronary syndrome, and successful percutaneous coronary intervention (PCI) were performed with intravascular ultrasound (IVUS) guidance.
2. Patients having coronary plaques (≧ 500 µm in thickness or % plaque of 20% or more at ≧ 5 mm distal or proximal to the previously treated area in the same branch of coronary artery.

Exclusion Criteria:

1. Patients with bypass graft or in-stent restenosis at the site of PCI.
2. Patients who received PCI in the past on the lesion where the evaluation of coronary plaque volume is planned.
3. Patients who had plaques in a non-culprit site and might receive PCI during the treatment period.
4. Patients receiving lipid-lowering drugs (statins, fibrates, probucol, nicotinic acid or cholesterol absorption inhibitors).
5. Patients with familial hypercholesterolemia.
6. Patients with cardiogenic shock.
7. Patients receiving cyclosporine.
8. Patients with any allergy to Ezetimibe.
9. Patients with hepatobiliary disorders.
10. Pregnant women, women suspected of being pregnant, or lactating women.
11. Patients with renal disorders or undergoing dialysis.
12. Patients who are ineligible in the opinion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
the percent change in coronary plaque volume, the percent change in integrated backscatter signal obtained by integrated backscatter IVUS | 9-11 months

SECONDARY OUTCOMES:
absolute change from baseline in coronary plaque volume, absolute and percent changes in minimal lumen diameter and percent stenosis, absolute and percent changes in total cholesterol and low-density lipoprotein cholesterol | 9-11 months

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Hibi, Principal Investigator — Yokohama City University Medical Center
Locations (1):
- Yokohama City University Medical Center, Yokohama, Kanagawa, Japan